CLINICAL TRIAL: NCT05112549
Title: Intrathecal Application of PD1 Antibody in Metastatic Solid Tumors With Leptomeningeal Disease (IT-PD1/ NOA 26)
Acronym: IT-PD1
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IT-PD1; 2021-001795-42 (EudraCT Number)
Record Dates: First submitted 2021-10-14; First posted 2021-11-09 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Leptomeningeal Disease
MeSH Terms: conditions — Meningeal Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Intervention Model Description: This is a single arm phase 1 trial with two parts.
  For part I (3+3 Design) there will be four cohorts:
  Cohort 1 with a fix dose of 20 mg, Cohort 2 with a fix dose of 30 mg, Cohort 3 with a fix dose of 40 mg and Cohort 4 with a fix dose of 50 mg.
  The dosage in the expansion part II will be fixe dosage for all patients depending on the results from Part I
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- intrathecal Nivolumab (Experimental): This is a prospective, interventional, open label, multicenter phase I trial in leptomeningeal disease in subjects with solid tumor that have a registered indication for intravenous treatment with PD1 antibody. Subject will undergo 6 cycles each 14 days in duration and a safety visit 7 days after the 3th dosage and 7 days after the 6th dosage. The Follow-up phase will start four weeks after the last dose and will continue monthly (up to 4 Follow-up visits in total).The study consists of two parts:
  Part I "dose - escalation phase" (3 + 3 design) with 4 cohorts and each subject will receive an intrathecal nivolumab treatment with a fixed predefined dose (20 mg, 30 mg, 40 mg or 50 mg). On each dose level, exposure of subjects to intrathecal nivolumab will follow a staggered approach. Part II "dose expansion phase": subjects will receive an intrathecal PD1 treatment with a fixe dose, depending on the results from Part I.
  Interventions: Drug: Nivolumab [Opdivo]

INTERVENTIONS:
Drug: Nivolumab [Opdivo] — Nivolumab (OPDIVO®) is a marketed pharmaceuticals material authorized in the European Union. This study uses an off-label route of administration of nivolumab. Subjects with leptomeningeal disease in solid tumours with an approved indication for intravenous treatment with the PD1 antibody will receive an intrathecal application of nivolumab. A total of six i.th. applications will be performed every 14 days. The intrathecal administration will be performed via an Ommaya reservoir or another intraventricular catheter.

SUMMARY:
To determine the safety of intrathecal (IT) PD1 antibody for Intrathecal application of PD1 antibody in metastatic solid tumors with leptomeningeal disease of solid tumors.

DETAILED DESCRIPTION:
Leptmeningeal disease (LMD) is an aggressive subtype of metastatic disease in the central nervous system (CNS) and has a poor prognosis with a median overall survival of a few months.The IT-PD1 trial group wants to contribute to an improvement of this situation for LMD patients by using an intrathecal application route for the PD1 antibody, i.e. a drug that has shown clinical efficacy in the underlying tumor via the intravenous route.

ELIGIBILITY:
Main Inclusion Criteria:

1. Patient aged ≥ 18 years at the time of signing the informed consent
2. Existing ability to understand and voluntarily sign an informed consent document prior to any study related assessments/procedures
3. Patient is at "good risk" ( NCCN guidelines version 1.2021)
4. Existence of the following Tumor board protocol confirmations: clinical recommendation for intrathecal therapy and evaluation of trial enrolment & statement on the potential necessity of additional systemic treatment of metastatic tumor outside the CNS
5. Existing ability to adhere to the study visit schedule and other protocol requirements
6. Existing agreement to refrain from donating blood while on study drug and for 30 days after discontinuation from this study treatment
7. Karnofsky performance score > 50%
8. Diagnosis of LMD by CSF and/or MRI (details see Study protocol)
9. If radiation therapy was performed please confirm: Participants eligible for IT-PD1 should have completed their radiation therapy due to clinical indication > 2 weeks prior to enrollment into the trial
10. Neurological examination (NANO scale) acc. Nayak et al., 2017 performed
11. MRI assessment at screening is based on the LANO scorecard acc. to Le Rhun et al., 2019
12. Existing ability to undergo intrathecal therapy via an intraventricular catheter (e.g. Ommaya reservoir)
13. Primary tumor tissue for the assessment of PD-1 and PD-L1 is optional at the timepoint of inclusion and enrollment but does need to be shipped before end of the trial.
14. Existing willingness of female patient of childbearing potential and male patient with female partner of childbearing potential to use highly effective contraceptive methods during treatment and for 150 days (male or female, see SmPC) after the last dose (details see Study protocol)

Main Exclusion Criteria:

1. Women during pregnancy and lactation.
2. Previous intrathecal nivolumab application.
3. Patient at "poor risk" (NCCN guidelines version 1.2021)
4. The following differential diagnoses to LMD are exclusion criteria: a. Aseptic, meningitis b. Viral meningitis, c. Bacterial meningitis
5. History of hypersensitivity to monoclonal antibodies
6. Participation in other clinical AMG or MDR trials or observation period of competing trials or if there is otherwise a high risk of insurance law issues intervening between two studies and if the participation affects the primary endpoint of the IT-PD1 study. In case of uncertainty, competing insurances must be contacted prior to participation
7. A clinical condition that in the opinion of the investigator would interfere with the evaluation or interpretation of patient safety or trial results or that would prohibit the understanding of informed consent and compliance with the requirements of the protocol
8. Any treatment-related toxicities from prior systemic anti-tumor or immune therapy not having resolved to CTCAE version 5.0 grade 1, with the exception of alopecia
9. Patient with confirmed history of current autoimmune disease
10. Patients with any disease resulting in permanent immunosuppression or requiring permanent immunosuppressive therapy
11. Existence of clinically significant active infection (details see study protocol)
12. Inability to undergo MRI with contrast agent
13. The underlying primary tumor has not a registered and authorized indication in the European Union for intravenous treatment with Nivolumab, Pembrolizumab or Atezolizumab (details see study protocol). In addition, leptomeningeal disease of solid tumors with a high tumor mutational burden is also eligible.
14. Existence of abnormal laboratory values for the following values in hematology, coagulation parameters, liver and renal function (details see study protocol)
15. Patients who have received live or attenuated vaccine therapy used for prevention of infectious disease within 4 weeks of the first IT application of nivolumab
16. Patients requiring chronic systemic corticosteroid therapy (> 10 mg prednisone or equivalent per day) or any other immunosuppressive therapies (including anti-TNF-a therapies)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2021-10-12 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of Adverse Events for Dose Limiting Toxicities [Safety and Tolerabillity] | up to 4 months after last dose
  This trial will investigate the maximum tolerable dose and safety of intrathecal PD1 antibody administration in LMD of metastatic solid tumors with a registered indication for treatment with intravenous PD1 antibody or PD-1L antibody. The safety endpoints will be assessed by a review of adverse events and serious adverse events according to CTCAE up to 4 months days after last dose.Subjects will undergo 6 cycles each 14 days in duration and a safety visit 7 days after the 3th dosage and 7 days after the 6th dosage.The appropriate dose for the expansion phase (Part II) is based on the results in Part I (dose escalation phase) and will define the maximum tolerable fix dose in Part II.

SECONDARY OUTCOMES:
Overall Survival | last follow-up, up to 4 months after last dose
  The secondary endpoint is overall survival defined as the time interval from the date of first study administration to the date of progression.

CONTACTS AND LOCATIONS:
Overall Officials: Ghazaleh Tabatabai, Prof.Dr., Study Director — University Hospital Tuebingen
Locations (9):
- Germany (9):
  - Universitätsklinikum Bonn, Bonn
  - University Hospital Freiburg, Neurosurgery, Freiburg im Breisgau
  - University Hospital Heidelberg, Neurooncology, Heidelberg
  - SLK-Kliniken Heilbronn GmbH Klinik, Heilbronn
  - University Hospital Mannheim, Neurology Clinic, Mannheim
  - Klinikum rechts der Isar/Technische Universität München, München
  - Katharinenhospital Stuttgart, Stuttgart
  - University Hospital Tübingen, Neurooncology, Tübingen
  - University Hospital Ulm, ECTU - Early Clinical Trail Unit, Ulm